CLINICAL TRIAL: NCT04354233
Title: A National, Multicenter, Randomized Controlled Trial to Assess the Efficacy of a Physical Activity Program to Improve Quality of Life and Reduce Fatigue in Women With Metastatic Breast Cancer
Brief Title: A Physical Activity Program to Improve Quality of Life and Reduce Fatigue in Metastatic Breast Cancer
Acronym: ABLE02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Fondation ARC (Other); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ABLE02; ET20-022 (Other: Sponsor ID)
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Physical activity; Connected devices; e-Health; Quality of life; Fatigue
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: At the first visit of the study, participants will be randomly assigned (1:1 ratio), with minimization based on the presence of visceral metastases (presence vs. absence of visceral metastases), the method of administration of chemotherapy (intravenous vs. per os) and the 6-minute walking distance (6MWD) (<455 versus ≥ 455m based on the median of the pilot ABLE study) to: (i) the intervention arm to receive PA recommendations and benefit from a 6-month APA program (ii) the control arm to receive PA recommendations only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention with connected devices (Experimental): Women randomized to the intervention arm will follow a 6-month physical activity intervention using a connected device that includes an activity tracker, a smartphone and a mobile application. Patients will also receive physical activity international recommendations
  Interventions: Device: Physical activity intervention with connected devices
- Standard care (No Intervention): Women will receive stardard care and physical activity international recommendations, without further intervention

INTERVENTIONS:
Device: Physical activity intervention with connected devices — Participants randomized in the intervention arm will receive recommandations in physical activity. They will also receive an activity tracker Withings Steel to wear during 6 months. The tracker will be connected to the "Withings Health Mate" application and the ABLE02 application. Participants will be encouraged to practice at least three walking sessions weekly of more than 10 consecutive minutes. Concerning the number of steps per day, the first objective will be determined according to the 6-min walking distance and to participants' preferences and capacities. The objective will be recalculated monthly according to the number of steps performed the previous week and will be adapted by the physical activity (PA) instructor and participants. Phone calls with the participants are regularly planned. Weekly quizzes on PA and nutrition will be proposed through the ABLE02 application. A messaging system and a phone line will be available for participants to contact the study team.
  Arms: Physical activity intervention with connected devices

SUMMARY:
INTRODUCTION: Patients with a metastatic breast cancer suffer from a deteriorated quality of life and numerous symptoms such as pain, severe fatigue and a decrease of their physical fitness. As the feasibility of a physical activity program has been demonstrated in this population, ABLE02 aims to assess the efficacy of a 6 month-physical activity program based on connected devices to improve health-related quality of life and to reduce fatigue in women with metastatic breast cancer.

METHODS/ANALYSIS: ABLE02 is a prospective, multicenter, randomized, controlled and, open-label study. 244 patients with a metastatic breast cancer , at least one positive hormone receptor and a first-line chemotherapy planned will be randomly assigned (1:1 ratio) to: (i) the intervention arm to receive physical activity recommendations, an activity tracker to wear 24 hours a day during the whole intervention (6 months) with at least three walking sessions weekly and quizzes to answer each week on physical activity and nutrition (ii) the control arm to receive physical activity recommendations only. Assessments will be conducted at baseline, M3, M6, M12 and M18 to evaluate the clinical, physical, biological and psychological parameters and survival of participants. All questionnaires will be completed on a dedicated application.

DISCUSSION: An activity program based on smartphone application linked to an activity tracker may help to improve quality of life and reduce fatigue of patients with a metastatic breast cancer. The growth of e-health offers the opportunity to get real-time data as well as improving patient empowerment in order to change long-term behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 1) female,
* 2) ≥ 18 years old,
* 3) histologically confirmed metastatic breast cancer, with at least one positive hormone receptor (HR+) and HER2-,
* 4) first-line chemotherapy planned (or until 1 month after the chemotherapy has started) with intravenous (Paclitaxel or Doxorubicin or Cyclophosphamide or Carboplatin) or per os (Capecitabine or Vinorelbine) administration - NB : a patient who has previously received one or more lines of hormone therapy and who must start a 1st line of chemotherapy is eligible,
* 5) Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2,
* 6) life expectancy ≥ 3 months,
* 7) willing to be involved throughout the study,
* 8) ability to practice a adapted physical activity (APA) certified by a medical certificate issued by the referring oncologist or the clinical investigator,
* 9) using a compatible smartphone or Tablet PC to download the application ABLE02 and Withings Health Mate (from iOS 10 and android 6.0 and more recent),
* 10) Internet access,
* 11) valid health insurance affiliation,
* 12) able to read, write and understand French.

Exclusion Criteria:

* 1) presence of unstable bone metastases or unconsolidated pathological fractures,
* 2) presence of central nervous system involvement with neurological deficits that prevent from walking,
* 3) presence of a history or co-existence of other primary cancer (except of in situ cancer regardless of the site and/or basal cell skin cancer and/or non-mammary cancer in complete remission for more than 5 years),
* 4) severe undernutrition (HAS) (i.e. for women ≤ 70 years old: a weight loss of ≥ 15% in 6 months or ≥10% in 1 month and for women over 70 years old: a weight loss of ≥ 15% in 6 months or ≥10% in 1 month, and body mass index <18 kg/m²),
* 5) presenting a PA contraindication (e.g., uncontrolled hypertension, uncontrolled heart disease),
* 6) concurrent participation in another PA study,
* 7) unable to be followed for medical, social, family, geographical or psychological reasons throughout the study,
* 8) deprived of liberty by judicial or administrative decision,
* 9) pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
time to deterioration of global health status (GHS) score of EORTC QLQ C30 | Month 18
  Health-Related Quality of Life (HRQoL) and fatigue will be measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ-C30). QLQ-C30 questionnaire consists of 30 items to evaluate 5 functioning domains (physical, role, emotional, cognitive, and social), a global HRQoL domain, 3 symptom domains (pain, fatigue and nausea) and 6 single items (dyspnea, insomnia, anorexia, diarrhea, constipation and financial impact). Participants will answer to a Likert scale ranging from "not at all" to "very much" and from "very bad" to "excellent" only for the global HRQoL questions. All scores will be standardized to a 0 to 100 scale according to the EORTC scoring manual. Higher scores represent better functioning, better global HRQoL and greater symptom burden.
  Deterioration is defined as a 5-point decrease relative to baseline in GHS score, with no subsequent increase above this threshold.
time to deterioration of fatigue score of EORTC QLQ C30 | Month 18
  Health-Related Quality of Life (HRQoL) and fatigue will be measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ-C30). QLQ-C30 questionnaire consists of 30 items to evaluate 5 functioning domains (physical, role, emotional, cognitive, and social), a global HRQoL domain, 3 symptom domains (pain, fatigue and nausea) and 6 single items (dyspnea, insomnia, anorexia, diarrhea, constipation and financial impact). Participants will answer to a Likert scale ranging from "not at all" to "very much" and from "very bad" to "excellent" only for the global HRQoL questions. All scores will be standardized to a 0 to 100 scale according to the EORTC scoring manual. Higher scores represent better functioning, better global HRQoL and greater symptom burden.
  A deterioration of fatigue is defined as a 5-point increase relative to baseline fatigue score, with no subsequent decrease above this threshold.

SECONDARY OUTCOMES:
Overall survival | Month 18
  Period from the date of randomization to the date of event defined as death from any cause
Progression free survival | Month 18
  Period from the date of randomization to the date of event defined as progression of the disease or death from any cause
Other dimensions of health-related quality of life of the EORTC QLQ C30 | Baseline, Month 3, Month 6, Month 12
  Health-Related Quality of Life (HRQoL) and fatigue will be measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ-C30). QLQ-C30 questionnaire consists of 30 items to evaluate 5 functioning domains (physical, role, emotional, cognitive, and social), a global HRQoL domain, 3 symptom domains (pain, fatigue and nausea) and 6 single items (dyspnea, insomnia, anorexia, diarrhea, constipation and financial impact). Participants will answer to a Likert scale ranging from "not at all" to "very much" and from "very bad" to "excellent" only for the global HRQoL questions. All scores will be standardized to a 0 to 100 scale according to the EORTC scoring manual. Higher scores represent better functioning, better global HRQoL and greater symptom burden.
  All of the secondary health-related quality of life dimensions except the global score and fatigue are evaluated.
Fatigue | Baseline, Month 3, Month 6, Month 12
  Multidimensional aspects of fatigue will be assessed by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-FA12 cancer related fatigue module. EORTC QLQ-FA12 consists of 12 items to evaluated physical, cognitive and emotional domains of cancer-related fatigue. Participants will answer to a 4-points Likert scale ranging from "not at all" to "very much". All scores will be transformed to a 0 to 100 scale and higher scores will indicate greater degree of fatigue.
Proportion of patients who change their physical condition (6-min walking distance) | Change between baseline, Month 3, Month 6 and Month 12
  6-min walking distance
Proportion of patients who change their physical condition (sit-to-stand) | Change between baseline, Month 3, Month 6 and Month 12
  Sit-to-stand
Proportion of patients who change their physical condition (handgrip strength) | Change between baseline, Month 3, Month 6 and Month 12
  Handgrip strength
Proportion of patients who change their weight | Change between baseline, Month 3, Month 6 and Month 12
  Body weight (kg)
Proportion of patients who change their waist circumference | Change between baseline, Month 3, Month 6 and Month 12
  Waist circumference (cm)
Proportion of patients who change their hip circumference | Change between baseline, Month 3, Month 6 and Month 12
  Hip circumference (cm)
Proportion of patients who change their physical activity level | Change between baseline, Month 3, Month 6 and Month 12
  PA level will be measured by the Godin Leisure-Time Exercise Questionnaire (GSLTPAQ). The GSLTPAQ is a short validated self-administrated physical activity (PA) questionnaire which includes three main questions about frequency of low (e.g., easy walking), moderate (e.g., brisk walking), and strenuous (e.g., jogging) leisure-time PA of at least 15 minutes duration in a typical week. The total score is obtained by multiplying frequencies from mild, moderate and strenuous PA by three, five and nine metabolic equivalents respectively and adding these together. Finally this score is divided into three categories (≥ 24 units is equivalent to mild active; between 14 and 23 units is equivalent to moderately active and < 14 units is equivalent to insufficiently active).
Proportion of patients who change sleep disorders | Change between baseline and Month 6
  Perceived sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI) evaluating seven sleep components: (1) sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbance, (6) use of sleeping medication, and (7) daytime dysfunction. Each of the seven components is rated on a Likert scale from "Not during last month" (0) to "3 or 4 times per week" (3). The total score resulting from the sum of the seven components ranges from 0 to 21, and a cut off 5 has been found to reflect clinically significant sleep disturbances.
  The quality of sleep will also be evaluated by the activity tracker based on automatic recognition of total duration of sleep, duration of deep and light sleep per night for the intervention arm only.
Proportion of patients who loss muscle mass (sarcopenia) | Change between baseline, Month 3, Month 6, Month 12 and at first progression up to Month 18
  CT scans
Proportion of patients who change their dietary patterns | Change between baseline and Month 6
  Dietary patterns will be assessed using a qualitative food frequency questionnaire composed of 35 items. Participants will answer the question "how frequently do you consume this product" on a Likert-type scale ranging from "never or almost" to "once per day or more" (stating quantity only for the range "once per day or more"). The questionnaire will characterize the consumption of fruits, vegetables, cereals, milk, dairy products, bread, meat, fish, poultry, eggs, starches, plant fat, desserts, sweetened products, non-alcoholic beverages, cold cuts, fried food, fast foods, preprepared meals, crackers, and snacking.
Proportion of patients who have severe toxicity (grade > 2) | Month 12
  Occurrence of severe toxicity (grade > 2) according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Proportion of patients who have modifications in inflammation and sarcopenia according to blood sample analysis | Change between baseline, Month 3, Month 6, Month 12 and at first progression up to Month 18
  Two 10mL blood samples will be collected before each physical assessment and before starting chemotherapy and at 1st progression.
  The following assays will be performed on plasma for the assessment of inflammation and biomarker of sarcopenia: Myostatin, Activin, Cortisol, TNF-alpha, IFN-gamma, IL-1beta, IL-6, Follistatin, GDF5 (BMP14), IL-10, IL-15, NH3, Aminogram.
  The levels of lymphocytes, monocytes, neutrophils will be extracted from the data of the routine blood test.
Proportion of patients who have modifications on oxidative stress according to blood sample analysis | Change between baseline, Month 3, Month 6, Month 12 and at first progression up to Month 18
  Two 10mL blood samples will be collected before each physical assessment and before starting chemotherapy and at 1st progression.
  The following assays will be performed on plasma for the assessment of oxidative stress: Advanced oxidation protein products (AOPP), malondialdehyde (MDA), Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX), Xanthine oxidase (XO), and Myeloperoxidase (MPO).
Proportion of patients who modify their personnality factors | Change between baseline and Month 6
  Based on the Five-Factor Model, personality traits will be assessed by the French Big Five Inventory questionnaire (BFI-Fr). The BFI-Fr contains 45 self-descriptive statements that assess the 5 personality traits: neuroticism (which refers to a propensity to experience negative emotions, distress, and anxiety), extraversion (a propensity to be energetic, sociable, and experience positive emotions); openness to experience (the tendency to be curious, imaginative, and to entertain new ideas, values, and experiences); conscientiousness (reflecting self-disciplined, planful, and organized); and agreeableness (which refers to cooperativeness and altruism). Each item was rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). All items will be recoded in the direction of the trait label, and the mean will be taken across items for each personality trait.
Proportion of patients who modify their behaviour in association with physical activity | Change between baseline and Month 6
  The process of change will be evaluated by a validated scale constructs from the transtheoretical model. The process of change scale is a 22-item self-administrated questionnaire to measure eight process of change: self-reevaluation (item 4,8 and 12), reinforcement management (items 7,15 and 12), self-liberation (items 8, 16 and 22), dramatic relief (items 2 and 10), environmental reevaluation (items 3 and 11), counterconditioning (items 5, 13 and 19), helping relationships (items 6, 14 and 20) and consciousness raising (items 1, 9 and 17). Participants will answer to a Likert scale ranging from 1 (never) to 5 (very often). Items in each process of change will be added and then an average score will be calculated. When the average is ≥ 3, the process of change is activated.
Proportion of patients who accept the connected device (in the intervention arm only) | Month 6
  Acceptability questionnaire will be assessed by a 21-item questionnaire to evaluate satisfaction concerning the use of connected devices (application, website, quizz, activity tracker).
Proportion of patients who are compliant to the PA intervention (in the intervention arm only) | Month 6
  Performed 3 PA sessions per week
Proportion of patients who modify their cognition | Change between baseline, Month 6 and Month 12
  The cancer-related cognitive impairment will be measured by the Functional Assessment of Cancer Therapy-Cognition (FACT-Cog). The FACT-Cog is a validated self-administrated questionnaire in order to assess memory, attention, concentration, language, and thinking abilities. The questionnaire is composed of 37 items with four subscales: patients' perceived cognitive impairments, perceived cognitive abilities, deficits observed or commented on by others, and impact of cognitive changes on HRQoL. Participant will answer how often this situation occurred during the last 7 days on a Likert-type scale ranging from "never" to "several times a day". For both scales, higher scores indicated better perceived cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier TREDAN, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - Institut de Cancérologie de l'Ouest (ICO), Angers
  - CHU Avignon, Avignon
  - CH Fleyriat, Bourg-en-Bresse
  - CH Cotentin, Cherbourg
  - CH Cholet, Cholet
  - CGFL, Dijon
  - Groupement Hospitalier Mutualiste, Grenoble
  - Centre Léon Bérard (CLB), Lyon
  - Hospices Civils de Lyon, Lyon
  - CH Morlaix, Morlaix
  - AP-HP, Paris
  - Institut Curie, Paris
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie Lucien Neuwirth (ICLN), Saint-Etienne
  - Institut de Cancérologie de l'Ouest (ICO), Saint-Herblain
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delrieu L, Anota A, Tredan O, Freyssenet D, Maire A, Canada B, Fournier B, Febvey-Combes O, Pilleul F, Bouhamama A, Caux C, Joly F, Fervers B, Pialoux V, Perol D, Perol O. Design and methods of a national, multicenter, randomized and controlled trial to assess the efficacy of a physical activity program to improve health-related quality of life and reduce fatigue in women with metastatic breast cancer: ABLE02 trial. BMC Cancer. 2020 Jul 3;20(1):622. doi: 10.1186/s12885-020-07093-9. PMID 32620149